CLINICAL TRIAL: NCT07191678
Title: Mechanisms Affecting the Gut of Preterm Infants Receiving Blood Transfusion With Different Enteral Feed Interventions
Acronym: MAGPIE-2
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: University of Leeds (Other); Imperial College London (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23HH8296
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: NEC - Necrotizing Enterocolitis; NEC; Preterm Babies; Preterm Infant Health
Keywords: NEC; Necrotizing Enterocolitis; Necrotising Enterocolitis; Preterm
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Withhold feeds during routine packed red cell transfusion: Infants who have been randomised in the WHEAT Trial to have their enteral feeds withheld during routine packed red cell transfusion.
- Continue feeds during routine packed red cell transfusion: Infants who have been randomised in the WHEAT Trial to have their enteral feeds continued during routine packed red cell transfusion.

SUMMARY:
MAGPIE-2 is a prospective observational study designed to investigate the physiological mechanisms linking blood transfusion and enteral feeding practices to gut perfusion and oxygenation in very preterm infants. The study is nested within the WHEAT International randomised controlled trial, which compares two standard care approaches: withholding versus continuing milk feeds during red blood cell transfusion. While WHEAT evaluates clinical outcomes such as necrotising enterocolitis (NEC), MAGPIE-2 focuses on the underlying physiological changes that may contribute to NEC development.

NEC is a serious gastrointestinal condition affecting approximately 10% of extremely preterm infants and is associated with high mortality and long-term neurodevelopmental impairment. Previous observational studies have suggested a temporal link between blood transfusion and NEC onset, particularly when feeds are continued during transfusion. However, the mechanisms remain poorly understood.

MAGPIE-2 will use non-invasive monitoring tools-near-infrared spectroscopy (NIRS) and Doppler ultrasound-to measure cerebral and splanchnic (gut) tissue oxygenation and superior mesenteric artery (SMA) blood flow. These measurements will be used to calculate the Splanchnic-Cerebral Oxygenation Ratio (SCOR), a validated marker of gut tissue perfusion and ischaemia. A reduction in SCOR may indicate compromised gut oxygenation, potentially contributing to NEC.

The study will recruit 270 infants (135 per arm) already enrolled in the WHEAT trial. Weekly measurements will be taken until 34 weeks corrected gestational age or discharge. Peri-transfusion monitoring includes continuous NIRS from 4 hours before to 4 hours after transfusion, and additional 2-hour recordings at approximately 24 and 48 hours post-transfusion. SMA Doppler assessments will be performed weekly.

Primary outcomes include changes in SCOR post-transfusion between the two feeding strategies. Secondary outcomes include changes in cerebral and splanchnic oxygenation, SMA blood flow velocities, and the impact of severe anaemia (pre-transfusion haemoglobin ≤80 g/L) on these parameters. The study also includes an assessment of inter-operator variability in Doppler measurements.

MAGPIE-2 aims to provide mechanistic insights that could inform safer transfusion and feeding practices in neonatal care, potentially reducing the incidence of NEC in this vulnerable population.

DETAILED DESCRIPTION:
MAGPIE-2 is a mechanistic observational study nested within the WHEAT International randomised controlled trial, which compares two standard neonatal care practices: withholding versus continuing enteral feeds during red blood cell transfusion in very preterm infants. While WHEAT evaluates clinical outcomes such as necrotising enterocolitis (NEC), MAGPIE-2 is designed to explore the physiological mechanisms that may underlie the development of NEC in this context.

NEC is a leading cause of morbidity and mortality in extremely preterm infants, with onset often temporally associated with blood transfusion. The pathophysiology is thought to involve gut ischaemia, inflammation, and impaired perfusion, but the precise mechanisms remain unclear. MAGPIE-2 addresses this gap by applying non-invasive monitoring techniques to assess gut and brain oxygenation and perfusion in infants undergoing transfusion.

The study will recruit 270 infants (135 per arm) already enrolled in the WHEAT trial. These infants will undergo weekly and peri-transfusion assessments using near-infrared spectroscopy (NIRS) and Doppler ultrasound. NIRS will measure cerebral and splanchnic (gut) tissue oxygenation, allowing calculation of the Splanchnic-Cerebral Oxygenation Ratio (SCOR), a validated marker of gut perfusion. Doppler ultrasound will assess blood flow in the superior mesenteric artery (SMA), which supplies the gut regions most vulnerable to NEC.

Measurements will be taken:

Weekly (2-hour NIRS and SMA Doppler) until 34 weeks corrected gestational age or discharge Peri-transfusion: continuous NIRS from 4 hours before to 4 hours after transfusion (12-hour window), and 2-hour recordings at approximately 24 and 48 hours post-transfusion The primary outcome is the relative change in SCOR post-transfusion between the two feeding strategies. Secondary outcomes include changes in cerebral and splanchnic oxygenation, SMA peak systolic and diastolic velocities, and the relationship between pre-transfusion haemoglobin levels and perfusion metrics. The study also includes an assessment of inter-operator variability in Doppler measurements and a mediation analysis to explore causal pathways.

MAGPIE-2 will use mixed-effects regression models to account for within-subject and within-centre variability, and propensity score weighting to adjust for selection bias. The study is powered to detect a 20% absolute difference in SCOR, which is considered clinically significant for identifying gut ischaemia.

By integrating physiological data with clinical trial design, MAGPIE-2 aims to provide mechanistic evidence to support safer transfusion and feeding practices in neonatal care. The findings may inform future guidelines and reduce the incidence of NEC in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Very preterm babies (born between 23 to <30 weeks of gestational age ) in the WHEAT International trial
* Written informed consent from parents

Exclusion Criteria:

* Babies who are deemed too unstable to perform the non-invasive monitoring and the ultrasound scan measurements by the attending clinical team
* Babies who have already developed Bells stage 2 NEC, had bowel surgery or congenital abdominal conditions such as congenital diaphragmatic hernia, gastroschisis and exomphalos

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will recruit 270 very preterm infants born between 23 and 30 weeks gestational age who are already enrolled in the WHEAT International trial. These infants are receiving care in neonatal units across the UK participating in WHEAT. MAGPIE-2 will include 135 infants in each arm of the WHEAT trial (feeds withheld vs continued during transfusion). All participants must have informed parental consent for additional non-invasive monitoring. The study population represents a high-risk group for necrotising enterocolitis (NEC), and the inclusion criteria align with the WHEAT trial to ensure consistency in clinical context and intervention exposure. Exclusion criteria include infants with pre-existing NEC, congenital abdominal anomalies, or those deemed clinically unstable for monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-11-03 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Splanchnic-Cerebral Oxygenation Ratio (SCOR) post-transfusion | Continuous from 4 hours pre-transfusion to 4 hours post-transfusion (12-hour window) for each transfusion received with WHEAT Trial intervention; plus additional weekly 2-hour recordings until 34 weeks corrected age or neonatal discharge.
  SCOR is calculated as the ratio of splanchnic (gut) to cerebral tissue oxygenation, measured using near-infrared spectroscopy (NIRS). A reduction in SCOR may indicate gut hypoperfusion or ischaemia. This outcome assesses the relative change in SCOR following blood transfusion in infants whose feeds were withheld versus continued.

SECONDARY OUTCOMES:
Change in Cerebral Oxygenation (crSO2) Post-Transfusion | Continuous from 4 hours pre-transfusion to 4 hours post-transfusion (12-hour window) for each transfusion received with WHEAT Trial intervention; plus additional weekly 2-hour recordings until 34 weeks corrected age or neonatal discharge.
  Measures cerebral tissue oxygenation using NIRS to assess impact of transfusion and feeding strategy.
Change in Splanchnic Oxygenation (srSO2) Post-Transfusion | Continuous from 4 hours pre-transfusion to 4 hours post-transfusion (12-hour window) for each transfusion received with WHEAT Trial intervention; plus additional weekly 2-hour recordings until 34 weeks corrected age or neonatal discharge.
  Measures gut tissue oxygenation using NIRS to evaluate perfusion changes post-transfusion.
Change in SMA Peak Systolic Velocity Post-Transfusion | Weekly Doppler ultrasound assessments until 34 weeks corrected age or neonatal discharge.
  Assesses SMA blood flow velocity using Doppler ultrasound to evaluate gut perfusion.
Change in SMA Diastolic Velocity Post-Transfusion | Weekly Doppler ultrasound assessments until 34 weeks corrected age or neonatal discharge.
  Measures SMA end-diastolic velocity to assess vascular resistance and perfusion.
Relationship Between Pre-Transfusion Haemoglobin and SCOR, crSO2, srSO2 | Continuous from 4 hours pre-transfusion to 4 hours post-transfusion (12-hour window) for each transfusion received with WHEAT Trial intervention; plus additional NIRS weekly 2-hour recordings until 34 weeks corrected age or neonatal discharge.
  Evaluates association between haemoglobin levels and tissue oxygenation in gut and brain.
Relationship Between Haemoglobin and SMA Doppler Parameters | Weekly Doppler ultrasound assessments until 34 weeks corrected age or neonatal discharge.
  Assesses correlation between haemoglobin levels and SMA blood flow velocities and indices.
Inter-Operator Variability in SMA Doppler Measurements | One-time assessment during weekly Doppler ultrasound in a subset of 35 infants across 7 centres.
  Assesses consistency between operators in measuring SMA velocities and indices using ICC.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Charlotte's & Chelsea Hospital, Neontal Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No